CLINICAL TRIAL: NCT03222193
Title: Efficacy Study of the Medical Device TRP Snorless™ in the Treatment of Snoring
Acronym: SCORED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongue Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRP-S-001
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Snoring
Keywords: Medical device; Retraining; Snoring; TRP; Tongue
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRP group (Experimental): Snoring subjects treated with the Tongue Right Positioner (TRP) medical device
  Interventions: Device: TRP

INTERVENTIONS:
Device: TRP — 3 months of TRP tongue retraining

SUMMARY:
The Tongue Right Positioner (TRP Snorless™) is a medical device designed to restore physiological tongue positions when functioning or at rest and increase tongue muscles tone. Patient wears TRP Snorless™ daily at least 5 hours during night. Published data suggested that TRP Snorless™ increases oropharynx diameter and nasal patency, favouring airflow in upper airways. Independently of patient's adherence to daily myofascial exercises, the TRP Snorless™ treatment should increase tongue muscles' tone and decrease the risk of snoring during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years and ≤ 65 years at the time of signing informed consent
* Listed as continuous snorer (snoring at least 4 nights/week)
* Answer "Extremely loud" or "very loud" to question 1 of SBPS at screening
* Answer "very severe" or "severe" to question 2 of SBPS at screening
* Answer "extremely" or "quite a bit" to question 3 of SBPS at screening
* Dated and signed informed consent
* BMI ≤ 35

Exclusion Criteria:

* Severe Mandibular retrognathia and micrognathia
* Narrow and deep palate (less than 3 cm wide)
* Lack of three consecutive teeth in the area of (15-16-17-18) or (25-26-27-28).
* Lingual or labial short frenulum (the tongue cannot reach the upper incisors when mouth can be opened for two fingers)
* Intolerable gag reflex
* Known nasal septal deviation
* Neck circumference > 46 cm
* Patient currently treated for OSA
* Patient with AHI≥30 events/hour or with AHI>15 and (SFI) Sleep Fragmentation Index > 20
* Patient currently treated for central sleep apnoea
* Addiction to alcoholic beverages (5 drinks per day per NIAAA)
* Under constant pharmacological treatment for depression, anxiety, chronic pain, insomnia
* Hypertrophy of tonsils
* Macroglossia
* Hypertrophy of uvula
* Primary gastroesophageal reflux
* Any other pathology preventing subject from complying with the protocol
* Subject with recent oropharyngeal surgery or likely during the study
* Mental inability, unwillingness or language barrier precluding adequate understanding of or compliance with study procedures
* Pregnancy
* Patient with severe Chronic Obstructive Pulmonary Disease
* Asthmatic patient under inhaled corticoid therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Snore Index | 3 months
  number of snores >36 dB per hour of sleep by BresoDx

SECONDARY OUTCOMES:
Mean sound of snoring/night | 3 months
  (dB), in supine, non-supine and both positions by BresoDx
Maximum sound of snoring/night | 3 months
  (dB), in supine, non-supine and both positions by BresoDx
Sleep time | 3 months
  Total sleep time (h), in supine, non-supine and both positions by BresoDx
Apnoea Hypopnea Index | 3 months
  (AHI) Number of apnea/hypopnea per hour of sleep, in supine, non-supine and both positions by BresoDx
Orofacial functional score (NOT-S questionnaire) | 3 months
  Using NOT-S questionnaire
Tongue Endurance score | 3 months
  Using IOPI medical device
Quality of sleep | 3 months
  Using Spiegel questionnaire
Comfort / Safety | 3 months
  Using homemade questionnaire relative to TRP snorless TM
Nasal patency | 3 months
  Measure of the Peak Nasal Inspiratory Flow by In-check PNIF meter
Treatment compliance | 3 months
  Using the The TheraMon® temperature micro sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinika Šustova 1930/2, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No